CLINICAL TRIAL: NCT01905618
Title: RCT for Smoking Cessation in 10 Medical Schools
Brief Title: Tobacco Treatment Medical Education in 10 Medical Schools
Acronym: MSQuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Judith Ockene, Professor of Medicine, Division Chief, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 13353; 5R01CA136888 (NIH)
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Tobacco Use Disorder; Smoking Cessation
Keywords: Medical Education; Tobacco Dependence Treatment; Physician Delivered Intervention
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi Modal Education (MME) (Experimental): Medical students in the medical schools randomized to the MME will receive four interventions during the course of their medical education. The four interventions/components are: 1) web-based curriculum on tobacco dependence treatment; 2)tobacco counseling role play; 3) preceptor training and teaching medical students, preceptor modeling the 5As, student observation, and student feedback; and 4)booster session.
  Interventions: Behavioral: Web-based curriculum on tobacco dependence treatment; Behavioral: Tobacco Counseling Role Play; Behavioral: Preceptor Training and Teaching Medical Students; Behavioral: Booster Session
- Traditional Education (TE) (No Intervention): Medical schools randomized to the Traditional Education (TE) will represent usual care and includes the current content and mode for tobacco teaching in the medical school.

INTERVENTIONS:
Behavioral: Web-based curriculum on tobacco dependence treatment — The University of Massachusetts Medical School's web-based course, "Basic Skills for Working with Smokers" was adapted for this Randomized Controlled Trial (RCT). The goal is to provide standardized information in the following core tobacco content areas: epidemiology of tobacco use, health consequences of tobacco use, nicotine dependence and withdrawal assessment, and provision of behavioral and pharmacotherapy tobacco treatment. The course is 3 hours in length and can be completed at the student's convenience. The dean and the course director at each medical school required that the first year medical students complete the web-based curriculum prior to the next component of the study, the role play.
  Other Names: 5 As; Smoking Cessation; Nicotine dependence; Physician Delivered Intervention; Pharmacotherapy
  Arms: Multi Modal Education (MME)
Behavioral: Tobacco Counseling Role Play — The goal of the role play is to provide each student with the opportunity to apply what he/she learned in the web-based curriculum (the 5 As and the physician delivered intervention approach). The one hour session begins with a video of a patient-centered counseling approach which incorporates the 5A intervention presented in the web-based course. This is followed by a 30 minute role play session including various scenarios with physician/patient interaction. Students role play either as physician, patient or observer for each scenario.
  Other Names: 5 As; Smoking Cessation; Physician-Delivered Intervention
  Arms: Multi Modal Education (MME)
Behavioral: Preceptor Training and Teaching Medical Students — The goal of this intervention is to train preceptors in the use of the 5As with their patients and to teach and motivate their medical students to use the 5As. The academic detailing approach is used to provide a standardized 30 to 45 minute group training session during the third year clerkship. All preceptors and medical students are encouraged to intervene with patients who smoke. Preceptors are encouraged to model the 5As, observe and give feedback to the medical student in its use. Study-tailored handouts are available for preceptors and students. This component is implemented with the study cohort in their third year of medical school.
  Other Names: Physician Delivered Intervention; 5As; Preceptor modeling 5 As; Preceptor observation; Preceptor feedback; Academic Detailing
  Arms: Multi Modal Education (MME)
Behavioral: Booster Session — The last component of the intervention, a small group booster session, occurs during the third year of medical school. A five minute video reviews the use of the 5As and patient-centered counseling strategies. Faculty facilitate a small group discussion after viewing the video.
  Other Names: 5 As; Physician Delivered Intervention; Tobacco Dependence Treatment; Smoking Cessation
  Arms: Multi Modal Education (MME)

SUMMARY:
This study compares two methods of teaching the 5As (Ask, Advise, Assess, Assist, Arrange) for tobacco dependence treatment to medical students: 1) traditional medical education (TE), and 2) multi-modal education (MME). The MME arm builds upon the traditional curriculum at the medical school by providing a web-based instructional program, a role play, preceptor training, and a booster session. The hypotheses are that MME will outperform TE on observed 5As counseling skills on the Objective Structured Clinical Exam (OSCE); and MME will outperform TE on self-reported 5As counseling skills.

DETAILED DESCRIPTION:
Ten medical schools are matched and then randomized, with 5 schools being randomized to MME and 5 schools to TE.

The primary aim of the study is to refine, implement, and evaluate whether a multi-modal educational (MME) approach is more effective than traditional educational (TE) approach for developing skill in the use of the 5As counseling steps for tobacco dependence treatment.

Multi-Modal Education(MME)Approach:

The MME approach includes: 1) a web-based course during the first-year of medical school; 2) a tobacco counseling role-play exercise; 3) training preceptors in the use of the 5As, preceptor observation of students in the use of 5As and providing instruction and feedback to students during a designated third-year clerkship rotation; and 4) a booster session provided during the third-year clerkship experience. These components are designed to enhance the interpersonal (e.g. 5As self-reported skill, tobacco treatment knowledge), intrapersonal (e.g. experiences observing 5As, experiences receiving 5As instruction), and organizational factors (e.g. clinic/system reminders) associated with optimal learning. This combination, primarily due to the web-based course/role play and preceptor facilitated teaching methods, is hypothesized to enhance medical students' 5As tobacco dependence treatment skills, compared to the TE approach.

Traditional Education (TE) Approach:

The TE approach represents "usual care" and includes the current content and method for tobacco teaching among medical schools. TE content typically includes knowledge in the basic science of tobacco use (e.g. health consequences of tobacco use and passive smoking), and the knowledge and practice of tobacco dependence treatment. All schools prior to randomization met the inclusion criteria that the curriculum devoted no more than four hours to tobacco.

The RCT's secondary aims address the potential impact of the interpersonal, intrapersonal, and organizational factors on tobacco dependence treatment counseling skills. The hypothesis is that these factors mediate the relationship between the MME curriculum approach and the primary outcome, observed 5As counseling skill, and that the MME approach will outperform the TE approach in each of these areas. This study also will assess the feasibility of implementing the MME across medical schools.

ELIGIBILITY:
Inclusion Criteria:

Medical schools must have:-at least 90 first year medical students

* third year OSCEs, willing to add a tobacco-related OSCE, and able to provide access to each student's OSCE
* a tobacco curriculum not exceeding a total of four hours over the four years
* the flexibility within their curriculum to add and adopt new tobacco cessation modules
* willing and able to require first year students to enroll in the web-based course and to award credit for its successful completion
* a curriculum that includes a third year Family Medicine or Internal Medicine Clerkship
* resources to allow web-based training and electronic contact with students
* the ability to allow first and third year medical students to be surveyed

Exclusion Criteria:

Medical schools are excluded if they do not have:

* at least 90 first year medical students
* a third year OSCE, and are not willing to add a tobacco-related OSCE or able to provide access to student OSCEs
* a tobacco curriculum of less than four hours over the four years
* the flexibility within their curriculum to add and adopt new tobacco cessation modules
* the capacity to require first year students to enroll in the web-based course and to award credit for successful completion of the course
* a curriculum that includes a third year Family Medicine or Internal Medicine Clerkship
* resources to allow web-based training and electronic contact with students
* the ability to allow first and third year medical students to be surveyed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Objective Structured Clinical Exam (OSCE) | Up to 2 years
  The primary outcome is the observed tobacco treatment 5As counseling skills as measured by the Objective Structured Clinical Examination (OSCE), the standard method for evaluating medical student skill level at all U.S. medical schools.

SECONDARY OUTCOMES:
A self-report survey instrument for tobacco treatment counseling skill level | Up to 3 years
  The secondary outcome is the self report survey completed by first year medical students and then the followup assessment when completing the third year of medical school. All followup assessments will be completed by October 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Judith K Ockene, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (13):
- United States (13):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Stanford University School of Medicine, Stanford, California
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - University of Iowa Carver College of Medicine, Iowa City, Iowa
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - University of Louisville School of Medicine, Louiville, Kentucky
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - Harvard School of Public Health, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Creighton University School of Medicine, Omaha, Nebraska
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Ockene JK, Hayes RB, Churchill LC, Crawford SL, Jolicoeur DG, Murray DM, Shoben AB, David SP, Ferguson KJ, Huggett KN, Adams M, Okuliar CA, Gross RL, Bass PF 3rd, Greenberg RB, Leone FT, Okuyemi KS, Rudy DW, Waugh JB, Geller AC. Teaching Medical Students to Help Patients Quit Smoking: Outcomes of a 10-School Randomized Controlled Trial. J Gen Intern Med. 2016 Feb;31(2):172-181. doi: 10.1007/s11606-015-3508-y. PMID 26391030